CLINICAL TRIAL: NCT03031171
Title: Community Engaged Colon Cancer Screening Patient Navigator Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California, Davis (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SB09/10-034; 8P20GM103440-11 (NIH)
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: ColoRectal Cancer
Keywords: community engagement, navigation, cancer screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigated: Screening patient navigation (Experimental): Clinic patients who received navigation
  Interventions: Behavioral: Screening patient navigation
- Non-Navigated (Active Comparator): Randomly matched sample of non-navigated clinic patients
  Interventions: Behavioral: Non-Navigated

INTERVENTIONS:
Behavioral: Screening patient navigation — The program offered assistance with scheduling, paperwork, arranging transportation, answering questions and providing education about screening and colorectal cancer.
  Arms: Navigated: Screening patient navigation
Behavioral: Non-Navigated — Randomly matched sample of non-navigated clinic patients
  Arms: Non-Navigated

SUMMARY:
The goal of the project is to increase colorectal cancer screening within the priority population of female and male adults age 50 to 85 in Northern Nevada. A successful community-based cancer patient navigator program will be modified in partnership with the community into a multi-level screening intervention.

DETAILED DESCRIPTION:
The goal of the project is to increase colorectal cancer screening within the priority population of female and male adults age 50 to 85 in Northern Nevada. A successful community-based cancer patient navigator program will be modified in partnership with the community into a multi-level screening intervention. A well-tested behavioral change theory (the health belief model; HBM) will guide the intervention and the relative efficacy of a) the theory's constructs and b) evidence-based intervention practices on increasing screening rates will be examined. Although increased screening rates are associated with program navigators, it is unclear which program components are related to the outcome. In addition, there is ambiguity surrounding a) the temporal impact of the HBM on cancer screening and b) the relationships among the model's constructs. A quasi-experimental time-series design will be used to evaluate the outcome objective of increased screening rates by comparing screening rates one year pre- and post-intervention and whether navigated patients are better prepared for screening than non-navigated patients. A minimum of 315 participants (to correspond with a power level of .80) in the navigator program will be surveyed on knowledge about colorectal cancer, and satisfaction with and usefulness of the program. The anticipated contribution of the project will be to increase community efficacy, colorectal cancer screening in the project area, and to reduce cancer morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Insurance, no history of colon cancer,

Exclusion Criteria:

* No experience of relevant GI symptoms

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Colonoscopy completion | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devereux, PhD, MPH, Principal Investigator — University of Nevada, Reno
Locations (1):
- Univeristy of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No